CLINICAL TRIAL: NCT02042495
Title: A Clinical Trial to Evaluate Endometrial Cancer Biomarker Changes Following Exposure to the Insulin Sensitizer Metformin
Brief Title: Endometrial Cancer Biomarker Changes Following Exposure to Metformin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not obtain Health Canda approval for drug use in reasonable time and moved onward to new trial
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Shannon Salvador, MD, MSc, FRCSC, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JGH-140111
Record Dates: First submitted 2014-01-12; First posted 2014-01-23 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): Metformin 500 mg PO TID from time of entry to study until scheduled surgical staging operation.
  In cases of unresolving side effects, the metformin will be dose reduced to metformin 500 mg PO BID with evaluation after 1 week followed by withdrawal from the study if side effects persist.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin
  Other Names: glucophage

SUMMARY:
The investigators will explore the chemopreventive role of metformin. The purpose of this study is to determine whether, among patients with endometrial cancer, treatment with the currently approved insulin sensitizing drug metformin increases or decreases pathway activation distal to the insulin receptor in endometrial cancer tissue. This is a phase IIa study of metformin to be used to the pre-operative period of women diagnosed with endometrial cancer by comparing their endometrial biopsy specimens taken at their initial visit and after 4-6 weeks of treatment of metformin on the day of their surgical staging.

DETAILED DESCRIPTION:
Aim 1 To determine whether, among patients with endometrial cancer, treatment with the currently approved insulin sensitizing drug metformin increases or decreases pathway activation distal to the insulin receptor in endometrial cancer tissue.

Aim II To compare specified biomarkers in each endometrial cancer patient before and after receiving metformin. Our goal is to compare the following biomarkers in each patient before and after metformin administration: Ki-67, TUNEL assay for apoptosis level, phosphor-AMPK, phosphor-IGF-1R, phosphor-IRS1, phospho-Akt, phospho-S6, phosphor-mTOR, pACC.

All patients diagnosed with endometrial cancer presenting to the Jewish General Hospital for surgical treatment will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of endometrial cancer based on an endometrial sampling though biopsy or dilatation and curettage
* Must be able to undergo appropriate surgical staging for endometrial cancer
* Must consent to be in the study and must have signed and dated an IRB-approved consent form conforming to government and institutional guidelines

Exclusion Criteria:

* Patients with a contraindication to receiving metformin treatment
* Patients with cognitive impairment
* Renal or hepatic functioning > 125% upper limit of normal
* Currently on medications for metabolic diseases, such as diabetes mellitus
* History of lactic acidosis
* Treatment with medications that may increase metformin levels: cationic drugs, e.g., digoxin, amiloride, procainamide, trimethoprim, vancomycin, triamterene, and morphine
* History of chronic alcohol abuse

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in phosphorylated-S6 | 4-6 weeks
  Paired-t test will be used to determine the effect of oral metformin on the phosphorylated-S6 in pre-treatment and post-treatment endometrial samples.

SECONDARY OUTCOMES:
Effects of metformin on activation pathways downstream of the insulin receptor in endometrial samples by testing Ki-67 | 4-6 weeks
  Additional biomarker tested:
  * Ki-67
Assess each patients insulin resistive state using the HOMA (homeostatic model assessment) index | 4-6 weeks
  Assess the effect of metformin on pre-treatment and post-treatment biomarkers in serum to determine the HOMA index
  * fasting IGF-I
  * fasting insulin
  * fasting IGFBP-1
  * fasting glucose levels
Effects of metformin on activation pathways downstream of the insulin receptor in endometrial samples by testing the TUNEL assay | 4-6 weeks
  Additional biomarker tested:
  * TUNEL assay for apoptosis level
Effects of metformin on activation pathways downstream of the insulin receptor in endometrial samples by testing phosphorylated AMPK | 4-6 weeks
  Additional biomarker tested:
  * phosphorylated-AMPK
Effects of metformin on activation pathways downstream of the insulin receptor in endometrial samples by testing phosphorylated IGF-1R | 4-6 weeks
  Additional biomarker tested:
  * phosphorylated-IGF-1R
Effects of metformin on activation pathways downstream of the insulin receptor in endometrial samples by testing phosphorylated insulin-receptor substrate protein 1 (phosphor-IRS1) | 4-6 weeks
  Additional biomarker tested:
  * phosphor-IRS1
Effects of metformin on activation pathways downstream of the insulin receptor in endometrial samples by testing phosphorylated-Akt | 4-6 weeks
  Additional biomarker tested:
  * phospho-Akt
Effects of metformin on activation pathways downstream of the insulin receptor in endometrial samples by testing phosphorylated mTOR | 4-6 weeks
  Additional biomarker tested:
  * phosphor-mTOR
Effects of metformin on activation pathways downstream of the insulin receptor in endometrial samples by testing phosphorylated acetyl-CoA carboxylase (pACC) | 4-6 weeks
  Additional biomarker tested:
  * pACC

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada